CLINICAL TRIAL: NCT01634711
Title: A Prospective and Consecutive Clinical Evaluation of Soft Tissue Regeneration's L-C Ligament® in Primary ACL Reconstruction
Brief Title: Clinical Evaluation of a Resorbable PLLA Implant for Regeneration of the Anterior Cruciate Ligament (ACL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Soft Tissue Regeneration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC 1033, Version 3.0
Record Dates: First submitted 2012-06-22; First posted 2012-07-06 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Complete Tear, Knee, Anterior Cruciate Ligament
Keywords: ACL; Anterior Cruciate Ligament; Ligament; Resorbable polymer; Knee ligament

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The L-C Ligament (Experimental): Soft Tissue Regeneration's L-C Ligament is an interventional device intended for ACL reconstruction surgery within 13 weeks of acute rupture of the ACL and no previous treatment. The L-C Ligament temporarily replaces the human anterior cruciate ligament (ACL) and provides a bioresorbable scaffold within and around which the native ACL will regenerate over time.
  Interventions: Device: L-C Ligament

INTERVENTIONS:
Device: L-C Ligament — The L-C Ligament is a bioresorbable, three-dimensional (3-D) braided scaffold made from poly L-lactic acid (PLLA) fiber. One device is used to replace the ACL. The L-C Ligament is an interventional device. The L-C Ligament is comprised of three regions: (1) The femoral tunnel attachment site, (2) The ligament region (intra-articular zone), and (3) The tibial tunnel attachment site. For several months after surgery, the L-C Ligament replaces the function of the ACL. During this time, ligament tissue regenerates within and around the L-C Ligament, which is slowly absorbed and replaced by the ACL.
  Other Names: L-C Ligament. PLLA Scaffold. 3-D Bradied PLLA Devcie.

SUMMARY:
The purpose of this study is to evaluate the safety of a resorbable polymer implant (Soft Tissue Regeneration's L-C Ligament) for replacement and regeneration of the anterior cruciate ligament (ACL). Approximately 15 patients at 2-3 different hospitals in Europe will participate in this study. The hypothesis of this study is that the L-C Ligament will successfully regenerate the ACL with clinical outcomes similar to or better than surgical intervention with auto graft tissue.

DETAILED DESCRIPTION:
Reconstruction of the ACL is currently recommended as the standard of care following an ACL tear or rupture. The ACL has poor healing potential and repair of the damaged tissue is rarely successful. The gold standard for reconstruction of the ACL is autograft tissue, with the patellar and hamstring tendons the most common. The limitations of autograft are donor site morbidity and pain, and potential damage of the remaining tissue at the harvest site. Other problems include a limited amount of tendon available for harvesting, unpredictable resorption characteristics, and increased recovery time. Allografts are tissues such as patellar, hamstring, and Achilles tendons obtained from cadavers. The advantages of surgery with allograft are less pain and scarring, decreased surgical time, and faster rehabilitation. However, allografts can transmit disease, may elicit an unfavorable immunogenic response, and incorporate slower than autograft. Also, allografts cannot be sterilized without damaging the tissue, leading to a choice between a risk of bacterial infection and decreased tensile strength and healing potential.

The proposed study is a prospective, consecutive, non-randomized, multicentre clinical trial conducted at up to five European sites, wherein 15 study subjects will undergo primary ACL reconstruction with the L-C Ligament. After screening procedures are completed, eligible study subjects who provide written informed consent will be enrolled in the study. Subjects will undergo preoperative clinical, MRI, and radiographic evaluations and undergo primary ACL reconstruction. Follow-up clinical evaluations will be performed post-op (range 1-8 weeks), 3 months (± 3 weeks), 6 months (± 3 weeks), 12 months (± 1 month), and 24 months (± 2 months) after surgery. Assessment of safety (i.e., assessment of adverse events and complications), pain, and clinical function as well as imaging will occur.

In accordance with a separate radiographic protocol, analysis and scoring of MRI images (pre-op, 1 and 2 years), radiographs (pre- and post- op), and a CT scan post-op and at 1-year will be undertaken by an independent radiologist who will be masked to the identities of the subjects and clinical investigators. Outcome measures for imaging include position of the bone tunnels and interference screws, indirect evidence of ligament tissue remodeling, and evidence of tunnel-widening. Evidence of OA will also be monitored. The Principal Investigator and Co-Investigators will ensure that complications observed on radiographs, MRI, and CT images are reported to their ethics committee and the sponsor.

The primary objective of this study is to evaluate the safety of the L-C Ligament in primary ACL reconstruction. Safety will be evaluated by the occurrence, frequency, and severity of intra- and post- operative complications; the primary end point is one year and follow-up wil be performed for a minimum of two years. Clinical function will be assessed with the IKDC-2000 Scale and functionality of the device at two years follow-up.

The secondary objectives of this study are to determine efficacy by objectively and subjectively measuring pain, function, and the results of image analyses of the L-C Ligament in primary ACL reconstruction. Objective measures include the Lachman test, the anterior drawer test, the KT-1000 Arthrometer, the pivot-shift test, and the single-leg hop test. Pre- and post- operative objective and subjective measures include the Tegner and Lysholm scales. Pre- and post- op radiographs, MRI images pre-op, and at 1 and 2 years, and post-op and 1-year CT scans will be analyzed for position of the bone tunnels and screws, indirect evidence of ligament tissue remodeling, and evidence of widening of the bone tunnels.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 45 years of age.
2. Males and females.
3. If female, for the 24 months post-operative, actively practicing a contraception method, or surgically sterilised or postmenopausal.
4. Acute unilateral ACL tear, or partial or complete tear of the ACL that occurred within 18 weeks of injury, and requires reconstruction of the ACL.
5. Passive flexion ≥ 120° and passive extension on the target knee is the same as the contralateral knee.
6. Patients with all types of lateral and/or medial meniscal tears which are repairable.
7. Medial Collateral Ligament (MCL) grade 2 or less. Potential Subject is able to provide informed consent and must sign the EC-approved Informed Consent Form.
8. Must be physically and mentally willing and able to comply with post-operative rehabilitation and routinely scheduled clinical, radiographic and rehabilitation follow up visits through 24 months.

Exclusion Criteria:

1. Prior ACL reconstruction or other surgical procedure on the affected (target) knee.
2. Chronic ACL injury; interventional surgery scheduled 18 weeks or more after ACL injury.
3. Professional athletes currently engaged in active sport
4. Prior fracture of the affected (target) leg
5. Previous or current ACL injury on contra-lateral leg.
6. Multi-ligament reconstruction.
7. Malalignment with varus thrust
8. Patient greater than 193 cm tall (6' 4").
9. The patient does not follow pre-operative rehabilitation.
10. Confirmed connective tissue disorder.
11. Signs of moderate to severe degenerative joint disease (Osteoarthritis)
12. Concomitant injuries to the knee or lower extremities requiring treatment, per surgeon's discretion.
13. Severe pain, swelling, or redness within 24 hours prior to surgery.
14. Complete or partial Post Cruciate Ligament (PCL) tear.
15. Any of the following: 1/3rd meniscal resection; complex double-bucket tear; partially repaired meniscal tears.
16. Patient requires treatment of articular cartilage on target leg
17. The patient is mentally compromised.
18. The patient has a neuromuscular disorder that would engender unacceptable risk of knee instability, prosthesis fixation failure, or complications in postoperative care.
19. The patient has a diagnosed systemic disease that would affect his/her safety or the study outcome.
20. The patient has an active or latent infection in or about the affected knee joint or an infection site distant from the knee that may spread to the knee hematogenously.
21. Pregnant based on a positive beta hCG serum or an in vitro diagnostic test result or breast-feeding.
22. The patient is obese with a BMI greater than or equal to 35.
23. The patient has a known allergy to PLLA.
24. The patient has a medical condition or comorbidity that would interfere with study participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
The anterior cruciate ligament (ACL) is clinically functional at one year follow-up | One year
  The primary outcome measure is that the ACL is functional one year postoperatively, and that no revision surgery was performed because of failure of the study device or loss of fixation directly attributable to the study device.

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) score | Pre-op, 6, 12, and 24 months
Tegner Activity score | Pre-op, 6, 12, & 24 months
Lachman test | Pre-op, 6, 12, and 24 months
KT-1000 Arthrometer score | Pre-op, 6, 12, 24 months
Lysholm Knee Score | pre-op, 6, 12, 24 months
Lachman Test score | pre-op, 6, 12, 24 months
Pivot Shift | pre-op, 6, 12, 24 months
Single-Leg Hop test | pre-op, 6, 12, 24 months
Anterior Drawer Test | pre-op, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Martini ziekenhuis, Groningen
  - Isala Klinieken - locatie Weezenlanden, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: For additional info and business inquries, visit www.softtissueregeneration.com or contact Joe Reilly, CEO, at jwreilly@softtissueregeneration.com — http://www.softtissueregeneration.com